CLINICAL TRIAL: NCT02345031
Title: A Balanced, Randomized, Placebo-Controlled, Double-Blind Study of the Efficacy and Safety of AUT00063 Versus Placebo in Age-Related Hearing Loss [CLARITY-1 Study]
Brief Title: Efficacy and Safety of AUT00063 Versus Placebo in Age-Related Hearing Loss
Acronym: CLARITY-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT022063
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Age-Related Hearing Loss
Keywords: hearing loss; speech-in-noise
MeSH Terms: conditions — Presbycusis; Hearing Loss | interventions — AUT00063

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AUT00063 (600 mg capsules) (Active Comparator): 3 capsules of 200 mg of the investigational drug AUT00063, to take orally once daily with food for 4 weeks
  Interventions: Drug: AUT00063
- (AUT00063 placebo capsules) (Placebo Comparator): 3 capsules of placebo, to take orally once daily with food for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUT00063 — 600 mg, orally, once a day, for 4 weeks
  Other Names: Experimental
  Arms: AUT00063 (600 mg capsules)
Drug: Placebo — orally, once a day, for 4 weeks
  Other Names: Comparator
  Arms: (AUT00063 placebo capsules)

SUMMARY:
This study aims to demonstrate that the investigational drug AUT00063 is effective and safe in the treatment of age-related hearing loss.

DETAILED DESCRIPTION:
Reduced activity at certain sites in the brain (called "voltage-gated potassium channels") has been linked to hearing problems, like age-related loss of hearing or tinnitus (a 'ringing' or buzzing noise in the ears).

AUT00063 is an experimental new medicine that enhances the action of these specific channels and so may treat the brain component of these hearing problems.

The main purpose of this study is to try to demonstrate an improvement in a speech-in-noise deficit after 4 weeks of treatment with the study drug versus the placebo (dummy drug which does not contain the drug). Subjects will undergo a safety follow-up after the treatment period.

Safety and efficacy will be determined by looking at a number of assessments (physical examinations, blood sampling, hearing assessments, questionnaires, etc.).

The amount of drug in the blood will also be measured. It is expected that around 70 people (at least 35 in each arm) with age-related hearing loss may take part in the study. The study participants will be recruited at around 13 sites in the USA.

ELIGIBILITY:
* Be between ages 50-89 years old
* American-English speaking
* Have difficulty hearing speech in a noisy environment
* No recent history of middle ear disease
* No severe insomnia, major depressive disorders, severe anxiety or post-traumatic stress disorder
* Not a current or previous user of hearing aids. You are eligible if you were noncompliant and stopped wearing a hearing aid device >6 months earlier for intermittent use or >3 years if you were a full-time consistent user of hearing aid devices
* Not be dependent on alcohol or drugs
* Have not participated in another research study within 30-days
* If female, you must confirm to be non child bearing (post-menopausal for at least 12-months or surgically sterile)
* If male, you must confirm to use a barrier method (condom)
* Not be a professional musician
* No history of important cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major disease deemed clinically significant by the study doctor

While you are in the study, you must:

* Follow the instructions you are given
* Come to the study centre for all visits with the study doctor or study staff
* Answer the telephone at the scheduled date and time for the 2 telephone calls
* Tell the study doctor or study staff about any changes in your health or the way you feel
* Tell the study doctor or study staff if you want to stop being in the study at any time
* Bring your Diary to each visit
* Not eat or drink anything containing Grapefruit beginning 7-days before Baseline visit (Visit 3, Day 1) until the end of the study
* Use sun screen if you plan to sunbathe
* Not use headphones or headsets at high volume
* Not use hearing aids or devices at any time during the study

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frisina, PhD, Principal Investigator — Director Global Center for Hearing and Speech Research
Locations (13):
- United States (13):
  - Sacramento ENT, Sacramento, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - ENT Associates of South Florida, Boca Raton, Florida
  - QPS MRA (Miami Research Associates), Miami, Florida
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - The University of Mississippi Medical Center, Jackson, Mississippi
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - PMG Research Inc., Wilmington, North Carolina
  - Piedmont Ear, Nose, & Throat Associates, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Jean Brown Research, Murray, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AUT00063 (600 mg Capsules) | (AUT00063 Placebo Capsules)
Started | 38 | 40
Completed | 37 | 39
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AUT00063 (600 mg Capsules) | (AUT00063 Placebo Capsules) | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants] — Population: Demographic data are listed from Full Analysis Set, excludes 2 subjects.
  Participants
    number analyzed (Participants) | 37 | 39 | 76
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 13 | 28
    >=65 years | 22 | 26 | 48
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics data are listed from Full Analysis Set, excludes 2 subjects
  Participants
    number analyzed (Participants) | 37 | 39 | 76
    Female | 15 | 17 | 32
    Male | 22 | 22 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographic data are listed from Full Analysis Set, excludes 2 subjects
  Participants
    Race: number analyzed (Participants) | 37 | 39 | 76
    Race: White/Caucasian | 36 | 38 | 74
    Race: Black/African-American | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographic data are listed from Full Analysis Set, excludes 2 subjects
  Participants
    Ethnicity: number analyzed (Participants) | 37 | 39 | 76
    Ethnicity: Hispanic Or Latino | 1 | 0 | 1
    Ethnicity: Not Hispanic Or Latino | 36 | 39 | 75
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 40 | 78
QuickSIN SNR-50 Score (dB) [Mean (Standard Deviation); unit: decibels (dB)] — The QuickSIN test measures the level of signal compared to the noise that is required to achieve 50% recognition and were administered in a sound booth at 70-dB HL binaurally. It is reported in decibels (dB). Population: QuickSIN data are listed from Full Analysis set, excludes 2 subjects
  decibels (dB)
    number analyzed (Participants) | 37 | 39 | 76
    (all) | 7.00 (1.963) | 7.11 (1.991) | 7.06 (1.965)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Loss After 4 Weeks of Treatment
Description: To compare the change in hearing using the QuickSIN test (speech in noise performance) from baseline (Day 1 to Day 28) between AUT00063 and placebo. The QuickSIN test measures the level of signal compared to the noise that is required to achieve 50% recognition. The test is administered in a sound booth at 70-dB HL binaurally via insert-ear phones. Three lists are administered to each individual subject and the threshold or 50% signal-to-noise ratio (SNR) is calculated as the mean of the three lists completed. Each list consists of six sentences with five key words to be scored per sentence. The sentences are presented in four-talker babble noise. The sentences are presented at pre-recorded signal-to-noise ratios which decrease in 5-dB steps from 25 (very easy) to 0 (extremely difficult).
Time Frame: 28 days
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: decibels (dB)
Arm/Group | AUT00063 (600 mg Capsules) | (AUT00063 Placebo Capsules)
Number analyzed (Participants) | 37 | 39
decibels (dB) | -1.114 [-1.956 to -0.272] | -1.914 [-2.703 to -1.125]

2. Secondary Outcome: Analysis of Change From Baseline in Adaptive Test of Temporal Resolution (ATTR) on End-Point Visit Day 28
Description: Final Average GDT Across-Channel at Day 28: Change from Baseline; FAS Population
Time Frame: 28 days
Population: FAS Population
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Arm/Group | AUT00063 (600 mg Capsules) | (AUT00063 Placebo Capsules)
Number analyzed (Participants) | 35 | 37
ms | -2.978 [-17.57 to 11.612] | -10.72 [-23.90 to 2.458]

3. Secondary Outcome: Analysis of Change From Baseline in Adaptive Test of Temporal Resolution (ATTR) on End-Point Visit Day 28
Description: Final Average GDT Within-Channel at Day 28: Change from Baseline; FAS Population
Time Frame: 28 days
Population: FAS Population
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Arm/Group | AUT00063 (600 mg Capsules) | (AUT00063 Placebo Capsules)
Number analyzed (Participants) | 36 | 39
ms | 4.452 [1.306 to 7.598] | 5.526 [2.661 to 8.392]

4. Secondary Outcome: To Further Investigate the Safety and Tolerability Profile of Repeat Administration of AUT00063 by Assessing Vital Signs, Physical Examination, Laboratory Exams and ECG
Description: Number of Subjects With At Least One Treatment Emergent Adverse Event
Time Frame: 42 Days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (AUT00063 Placebo Capsules): 3 capsules of placebo, to take orally once daily with food for 4 weeks
  Placebo: orally, once a day, for 4 weeks
Arm/Group | AUT00063 (600 mg Capsules) | Placebo (AUT00063 Placebo Capsules)
Number analyzed (Participants) | 38 | 40
Participants | 23 | 24

5. Secondary Outcome: Pharmacokinetic of AUT00063, Plasma Levels
Description: Exposure of AUT00063 ng/ml, in plasma levels at Day 28
Time Frame: 28 Days
Measure: Mean (Standard Deviation); unit: ng
Groups:
- Placebo: 3 capsules of placebo, to take orally once daily with food for 4 weeks
  Placebo: orally, once a day, for 4 weeks
Arm/Group | AUT00063 (600 mg Capsules) | Placebo
Number analyzed (Participants) | 36 | 36
ng | 3470.61 (1290.679) | 0 (0)

ADVERSE EVENTS:
Time Frame: The recording period for Adverse Events is the period starting from the Informed Consent signature until the safety close out visit or subject's study participation ends; a total duration of up to 10 weeks.
Arm/Group | AUT00063 (600 mg Capsules) | Placebo (AUT00063 Placebo Capsules)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/40
Other Adverse Events (participants affected / at risk) | 18/38 | 21/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUT00063 (600 mg Capsules) (N=38) | Placebo (AUT00063 Placebo Capsules) (N=40)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Acute Alcohol Intoxication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AUT00063 (600 mg Capsules) (N=38) | Placebo (AUT00063 Placebo Capsules) (N=40)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 — Back Pain
Blood triglycerides increased (Investigations) | 2 | 0 — Triglycerides increased
Diarrhoea (Gastrointestinal disorders) | 3 | 2 — Diarrhoea
Dizziness (Nervous system disorders) | 6 | 1 — Dizziness
Fatigue (General disorders) | 2 | 0 — Fatigue
Gastroenteritis (Infections and infestations) | 0 | 2 — Gastroenteritis
Headache (Nervous system disorders) | 4 | 5 — Headache
Nausea (Gastrointestinal disorders) | 2 | 3 — Nausea
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 — Sinus Congestion
Somnolence (Nervous system disorders) | 3 | 0 — Drowsiness
Tinnitus (Ear and labyrinth disorders) | 4 | 3 — Tinnitus
Upper respiratory tract infection (Infections and infestations) | 3 | 2 — Upper respiratory tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less